CLINICAL TRIAL: NCT00488306
Title: A Multicenter, Open Label Study to Evaluate the Efficacy and Safety of Tigecycline to Treat Complicated Intra-Abdominal Infections (cIAI) in Hospitalized Patients
Brief Title: Study Evaluating the Safety and Efficacy of Tigecycline in Hospitalized Patients With cIAI
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3074A1-101994
Record Dates: First submitted 2007-06-18; First posted 2007-06-20 (Estimated); Last update posted 2009-07-07 (Estimated); Status verified 2009-07

CONDITIONS: Abdominal Abscess
Keywords: Tigecycline; Complicated intra-abdominal infections; cIAI
MeSH Terms: conditions — Abdominal Abscess | interventions — Tigecycline

INTERVENTIONS:
Drug: tigecycline

SUMMARY:
In light of tigecycline's activity against these resistant bacteria, tigecycline may represent a viable new therapy for complicated intra-abdominal infections.

DETAILED DESCRIPTION:
To evaluate the efficacy and safety of tigecycline to treat complicated intra-abdominal infections in hospitalized patients. Both the clinical response profile and the microbiological response profile will be assessed. The primary endpoint will be clinical response within the microbiological evaluable population at the test-of-cure assessment.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized male or female patients greater than or equal to 18 years of age.
* Patients must be a candidate for or have had a laparotomy, or laparoscopy of an intra-abdominal abscess.
* Patients with a complicated intra-abdominal infection such as:

  * an intra-abdominal abscess;
  * an intra-abdominal abscess (including liver and spleen) that develops in a post-operative patient after receiving > 48 hours and less than or equal to 5 days of a non-study antibiotic. An intra-abdominal culture must be obtained from the infected site.
  * appendicitis complicated by perforation (grossly visible) and abscess and/or periappendiceal abscess;
  * perforated diverticulitis complicated by abscess formation or fecal contamination;
  * complicated cholecystitis with evidence of perforation or empyema;
  * perforation of the large or small intestine with abscess, or fecal contamination;
  * purulent peritonitis or peritonitis associated with fecal contamination;
  * gastric or duodenal ulcer perforation with symptoms lasting at least 24 hours prior to operation;
  * traumatic bowel perforation with symptoms lasting at least 12 hours prior to operation.

Exclusion Criteria:

* Patients with any concomitant condition that, in the opinion of the investigator, would preclude an evaluation of a response or make it unlikely that the contemplated course of therapy or follow-up visits could be completed.
* Active or treated leukemia or systemic malignancy that required treatment with chemotherapy, immunotherapy, radiation therapy or antineoplastic therapy within the past 3 months, or any metastatic malignancy to the abdomen with life expectancy less than 6 months.
* Anticipated length of antibiotic therapy less than 5 days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2006-08; Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
The primary efficacy endpoint will be clinical response within the clinically evaluable population at the test-of-cure assessment.

SECONDARY OUTCOMES:
microbiological response (eradicated, persistence, superinfection, or indeterminate) at the patient level, microbiological response (eradicated, persistence, or indeterminate) at the pathogen level (overall and resistant pathogens) clinical

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer; Trial Manager, Principal Investigator — For Taiwan, medinfo@wyeth.com
Locations (1):
- Multiple Cities, Taiwan